CLINICAL TRIAL: NCT05176145
Title: Demonstration of the Medical Interest of the VisioCyt® Artificial Intelligence Test
Acronym: DMIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vitadx (Other)
Collaborators: FONDATION FORCE POUR L'INNOVATION ET LA RECHERCHE EN SANTE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMIA-2021
Record Dates: First submitted 2021-12-03; First posted 2022-01-04 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Non-muscle Invasive Bladder Cancer (NMIBC)
Keywords: NMIBC; recurrence
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): Only one arm. The urine collection from each patient will be used for VisioCyt® test and conventional cytology
  Interventions: Device: VisioCyt®

INTERVENTIONS:
Device: VisioCyt® — * Cytological and endoscopic examination is planned as part of the usual management of patients under surveillance of Non-muscle invasive bladder cancer (NMIBC), according to the CCAFU guidelines.
  * Urine collection for conventional cytology and VisioCyt® test

SUMMARY:
European, multicenter clinical trial with VisioCyt®, an in vitro diagnostic medical device. VisioCyt® is an innovative solution for the early diagnosis of bladder cancer.

DETAILED DESCRIPTION:
VisioCyt® is based on a patented technology, combining bright-field imaging and artificial intelligence, from a simple urine sample from which the cells are extracted .

The main objective of the study is to demonstrate the medical superiority of the VisioCyt® test versus conventional cytology for detecting recurrence of bladder tumors, in patients monitoring non-muscle infiltrating bladder tumors at high and very high risk of progression

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and autonomous
* Patient understanding national language well and able to understand the protocol.
* Patient information and informed consent signature before the start of the study
* Patients under surveillance of Non-muscle invasive bladder cancer (NMIBC) at high and very high risk of progression, whatever the stage on the basis of a histological result. The diagnosis (primary or recurrence) should be less than or equal to 24 months (the last histology result confirming a bladder cancer with high or very high risk of recurrence is taken into account).

Exclusion Criteria:

* Patients who have had total bladder resection or bladder reconstruction
* Age <18 years old
* Person deprived of liberty or under guardianship (including curatorship)
* Bladder cancer outside of urothelial carcinoma
* Associated high urinary tract carcinoma
* Kidney transplant patient (BK virus)
* Pelvic radiotherapy patient (prostate cancer)
* Patients with or under surveillance of a muscle-infiltrating bladder tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Performance of VisioCyt® test vs conventional cytology | 24 months
  Sensibility of the cytological examination of urine with the VisioCyt® test and conventional cytology, all grades and stages combined

SECONDARY OUTCOMES:
Specificity, positive and negative predictive value for VisioCyt® test and conventional cytology | 24 months
  Specificity of the cytological examination of urine with the VisioCyt® test and conventional cytology, all grades and stages combined

CONTACTS AND LOCATIONS:
Locations (15):
- Hôpital Académique ERASME, Anderlecht, Belgium
- France (13):
  - CHU Angers, Angers
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Nantes, Nantes
  - Hôpital Bichat-Claude Bernard,, Paris
  - Hôpital Pitié-Salpétrière, APHP, Paris
  - Clinique la Croix du Sud, Quint-Fonsegrives
  - CHU de Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
- Pr Maria Jose Ribal, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No